CLINICAL TRIAL: NCT05473624
Title: A Phase I, Open-label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HRS-1167 as Monotherapy in Patients With Advanced Solid Tumors
Brief Title: Study of HRS-1167 as Monotherapy in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1167-I-101
Record Dates: First submitted 2022-07-13; First posted 2022-07-26 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-1167 (Experimental)
  Interventions: Drug: HRS-1167

INTERVENTIONS:
Drug: HRS-1167 — Participants will receive HRS-1167.

SUMMARY:
This study is designed to determine if treatment with HRS-1167 alone is safe, tolerable, and has anti-cancer activity in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18；
2. ECOG performance status 0-1;
3. Life expectancy is not less than 12 weeks;
4. Dose escalation and PK expansion part: Subjects diagnosed with advanced solid malignancies who are refractory to standard therapies or for which no standard therapy exists；
5. Efficacy expansion part：Ovarian Cancer、Breast Cancer、Pancreatic Cancer、Prostate Cancer or other cancer types with HRR gene mutation；
6. At least one target lesion (except maintenance therapy);
7. Adequate organ and marrow function as defined by the protocol.

Exclusion Criteria:

1. Surgery or chemotherapy within 4 weeks of the first dose of study treatment；
2. Subjects that are unable to swallow, or dysfunction of gastrointestinal absorption；
3. Active HBV/HCV/HIV infection;
4. Untreated and/or uncontrolled brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) of HRS-1167 | up to 24 days
Maximum tolerated dose (MTD) of HRS-1167 | up to 24 months
Recommended Phase II Dose (RP2D) of HRS-1167 | up to 24 months
AEs+SAEs | up to 24 months
  from the first drug administration to within 30 days for the last treatment dose

SECONDARY OUTCOMES:
Evaluation of pharmacokinetic parameter of HRS-1167: Cmax | At Cycle 0 Day 1, Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, and Cycle 4 Day 1 (each cycle is 21 days)
  The concentration of HRS-1167 in plasma will be determined (Cmax will be derived).
Evaluation of pharmacokinetic parameter of HRS-1167: Tmax | At Cycle 0 Day 1, Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, and Cycle 4 Day 1 (each cycle is 21 days)
  The concentration of HRS-1167 in plasma will be determined (Tmax will be derived).
Evaluation of pharmacokinetic parameter of HRS-1167: AUC | At Cycle 0 Day 1, Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, and Cycle 4 Day 1 (each cycle is 21 days)
  The concentration of HRS-1167 in plasma will be determined. Area under the curve is the integral of the concentration-time curve. The AUC reflects the actual body exposure to drug after administration. The AUC is dependent on the rate of elimination of the drug from the body and the dose administered.
Objective Response Rate (ORR) | up to 24 months
  Complete response + Partial response (CR+PR) based on RECIST 1.1.
Disease control rate (DCR) | up to 24 months
  Complete response + Partial response + Stable disease (CR+PR+SD) based on RECIST 1.1.
Duration of response (DoR) | up to 24 months
  Time from documentation of tumor response to disease progression assessed among patients who had an objective response.
Progression Free Survival (PFS) | up to 24 months
  Time from C1D1 to first assessment of disease progression or death, whichever is earlier.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Guangxi Medical University Affiliated Tumor Hosipital, Nanning, Guangxi
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shangdong
  - Shandong Cancer Hospital, Jinan, Shangdong
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhengjiang

IPD SHARING:
Plan to Share IPD: Undecided